CLINICAL TRIAL: NCT01428401
Title: Astragalus Membranaceus for Brain Edema Induced by Hemorrhagic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMR96-IRB-126
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Stroke; Hemorrhagic Transformation Due to Acute Stroke
Keywords: Complementary therapies; Acute hemorrhagic stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Chinese Herb Astragalus membranaceus
- Arm B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Chinese Herb Astragalus membranaceus — Astragalus membranaceus ( AM) at a rate of 3 g three times per day
  Arms: Arm A
Other: Placebo — at a rate of 3 g three times per day
  Arms: Arm B

SUMMARY:
Astragalus membranaceus (AM) is used to treat stroke for a long period, and a number of studies have known that AM can reduce cerebral infarction area and has anti-oxidation. Hemorrhagic stroke will induce secondary peri-blood clot edema and that may increase intracranial pressure to exacerbate clinical symptom. Therefore, the purpose of the present study was to investigate the effect of AM on hemorrhagic stroke edema. The investigators selected 80 hemorrhagic stroke patients , and who the stroke is first attack, they were randomly divided into control and experimental groups, and each group was 40 patients as follows: 1) control group, accepted AM placebo 2.8 g three times per day (tid) treatment for continuously 14 days from second day of admission or operation, except standard ordinary treatment; 2) experimental group, accepted AM 2.8 g tid treatment for continuously 14 days from second day of admission or operation, except standard ordinary treatment. Computer tomography (CT) examination was done at first day, 4th day and 7th day of admission, respectively. The ratio of brain edema was calculated by CT image, and inflammatory index including the levels of C-reactive protein (CRP), erythrocyte sedimentation rate (ESR)，Creatine Kinase BB Isoenzyme (CMBB). D-dimer from venous blood also were measured. In addition, the score including Glasgow outcome scale (GOS), Modified rankin scale (MRS), Function independence measure (FIM), Barthel index (BI) was recorded one week, four weeks and 12 weeks after admission or surgical operation, as an index for clinical symptoms. The index for the therapeutic effect of AM was according to above-mentioned the ratio of brain edema, inflammatory index and clinical symptoms.

The investigators expected the results of the present study may provide a scientific evidence for the hemorrhagic stroke edema treatment of AM, thus, the present study may contribute to use the method of integrated Chinese and Western Medicine for the treatment of stroke, and to the research of Chinese Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. female or male;
2. aged between 30 and 75 years;
3. randomized allocation to a study group within 24 hours of hemorrhagic stroke onset;
4. this was the patient's first hemorrhagic stroke, and the location of hemorrhage was the putamen;
5. treatment may or may not have been included surgery; and
6. the subject or their legal representative gave written informed consent to participate.

Exclusion Criteria:

1. recent thrombolysis treatment;
2. history of previous stroke;
3. full-dose or long-term anti-coagulation therapy;
4. hemorrhagic stroke but the location was not putamen;
5. coexisting systemic diseases such as terminal cancer, renal failure, liver cirrhosis, severe dementia, or psychosis;
6. participation in another clinical trial within the last three months; and
7. pregnancy or lactation.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
patients' scores(BI,FIM,GOS,mRS) on several clinical scales | baseline (within 7 ± 1 days after the onset of stroke) and week 4 (28 ± 4 days), and between at baseline and week 12 (84 ± 10 days).
  The primary outcome measures were the differences in patients' scores on several clinical scales, between baseline (within 7 ± 1 days after the onset of stroke) and week 4 (28 ± 4 days), and between at baseline and week 12 (84 ± 10 days). The scales we used were the Functional Independence Measure scale (FIM), Barthel Index scale (BI), Glasgow Outcome Scale (GOS), and Modified Rankin Scale (MRS). The scores of FIM, BI, GOS, and MRS were assessed by an experienced research nurse.

SECONDARY OUTCOMES:
inflammatory index and Computer tomography (CT) examination | at baseline (prior to the first AM dose), and again on the fourth and seventh day of admission
  1. inflammatory index, which included the levels of C-reactive protein (CRP) and erythrocyte sediment rate (ESR) for venous blood; these were measured at baseline (prior to the first AM dose), and again on the fourth and seventh day of admission; and
  2. Computer tomography (CT) examination, which was done at baseline and on the fourth and seventh days of admission. The ratio of brain edema was calculated by CT (volume of edema divided by blood clot volume)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chung Chen, master, Principal Investigator — d6407@mail.cmuh.org.tw